CLINICAL TRIAL: NCT00282698
Title: Outcomes With Use Of Intensive Insulin Therapy In Intraoperative Management Of Hyperglycemia In Adult Patients Undergoing Cardiac Surgery
Brief Title: Outcomes With Tight Control of Hyperglycemia in Cardiac Surgery Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 322-04
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Cardiac Surgical Procedures; Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

INTERVENTIONS:
Drug: Insulin infusion with a goal

SUMMARY:
Patients with or without diabetes may have high blood sugar levels due to stress response of the body during heart surgery. This study is being done to determine if maintaining normal blood sugar levels during open-heart surgery by using intravenous insulin results in a lesser incidence of death, wound infections in the chest, disturbances of heart rhythm, kidney failure, stroke and prolonged time on the breathing machine (artificial ventilation) within 30 days after surgery.

DETAILED DESCRIPTION:
Rigorous intraoperative glycemic control may be of paramount importance in affecting outcomes after cardiac surgery. There is evidence that strict control of glucose levels postoperatively results in improved outcomes in patients undergoing cardiac surgery. There is currently no consensus on optimal management of hyperglycemia intraoperatively. The aim of this prospective randomized controlled clinical trial is to determine whether normalization of intraoperative glucose levels with insulin improves outcomes. The comparison group will be treated with current standard practice to control hyperglycemia during surgery. The primary outcome is a composite of mortality, sternal wound infections, prolonged pulmonary ventilation, cardiac arrhythmias (new-onset atrial fibrillation, heart block requiring permanent pacemaker, cardiac arrest), stroke and acute or worsening renal failure within 30 days after surgery. Secondary outcome measures are length of intensive care unit and hospital stay as well as safety and efficacy of the study insulin infusion protocol.

ELIGIBILITY:
Inclusion Criteria

All subjects accepted for this study must be:

1. >=18 years of age
2. Undergoing an elective cardiac surgical procedure

Exclusion Criteria

Subjects who have one or more of the following will be excluded from the study:

1. Undergoing surgery not utilizing cardiopulmonary bypass
2. Unable to grant informed consent or comply with study procedure
3. Undergoing emergency open heart-surgery

3. Are allergic to any of the excipients in insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-07; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Mortality
Sternal wound infections
Stroke
Cardiac arrhythmias
Renal failure

SECONDARY OUTCOMES:
Lenght of intensive care unit stay
Length of hospital stay
Safety of study insulin infusion
Efficacy of study insulin infusion

CONTACTS AND LOCATIONS:
Overall Officials: Gunjan Y. Gandhi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Gandhi GY, Nuttall GA, Abel MD, Mullany CJ, Schaff HV, O'Brien PC, Johnson MG, Williams AR, Cutshall SM, Mundy LM, Rizza RA, McMahon MM. Intensive intraoperative insulin therapy versus conventional glucose management during cardiac surgery: a randomized trial. Ann Intern Med. 2007 Feb 20;146(4):233-43. doi: 10.7326/0003-4819-146-4-200702200-00002. PMID 17310047